CLINICAL TRIAL: NCT01206972
Title: Randomized, Double-blind, Parallel-group, Active-controlled, Dose-confirmatory Bridging Study of Rivaroxaban (BAY59-7939) 5 to 10 mg Once-daily Regimen With a Reference Drug of Enoxaparin in the Prevention of Venous Thromboembolism in Patients Undergoing Elective Total Knee Replacement
Brief Title: Dose-confirmatory Bridging Study in Total Knee Replacement
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 14398
Record Dates: First submitted 2010-09-20; First posted 2010-09-22 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Venous Thromboembolism
Keywords: venous thromboembolism; prevention; orthopaedic surgery
MeSH Terms: conditions — Venous Thromboembolism | interventions — Rivaroxaban; Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Experimental)
  Interventions: Drug: Rivaroxaban (BAY59-7939)
- Arm 2 (Experimental)
  Interventions: Drug: Rivaroxaban (BAY59-7939)
- Arm 3 (Experimental)
  Interventions: Drug: Rivaroxaban (BAY59-7939)
- Arm 4 (Active Comparator)
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Rivaroxaban (BAY59-7939) — daily dose: 5mg/day (5mg, once daily) for 11 to 12 days (±2 days)
  Arms: Arm 1
Drug: Rivaroxaban (BAY59-7939) — daily dose: 7.5mg/day (7.5mg, once daily) for 11 to 12 days (±2 days)
  Arms: Arm 2
Drug: Rivaroxaban (BAY59-7939) — daily dose: 10mg/day (10mg, once daily) for 11 to 12 days (±2 days)
  Arms: Arm 3
Drug: Enoxaparin — daily dose: 40mg/day (20mg, twice daily) for 10 to 11 days (±2 days)
  Arms: Arm 4

SUMMARY:
The objective of this dose-confirmatory bridging study is to investigate the safety and efficacy of rivaroxaban 5 to 10 mg once-daily (od) dosing in the prevention of venous thromboembolism (VTE) in Japanese patients undergoing elective total knee replacement (TKR) and to confirm the extrapolability of global data to Japanese patients by comparing with data from overseas phase III study (RECORD 3 - Study 11356) and phase II studies.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 20 years or above
* Patients undergoing elective TKR (the first replacement of the applicable knee joint)
* Patients' written informed consent to participation after receiving detailed verbal and written information on any study specific procedures in advance

Exclusion Criteria:

* Planned, staged major orthopedic surgery within 3 months prior to elective TKR or during this study
* History of clinically significant active bleeding (e.g. intracranial bleeding, gastrointestinal bleeding*), or high bleeding risk

  *: within 3 months prior to elective TKR for gastrointestinal bleeding
* Subjects with hepatic disease which is associated with coagulopathy leading to a clinically relevant bleeding risk
* Severe impaired renal function (CLCR calculated by Cockcroft-Gault formula: <30 mL/min)
* Conditions prohibiting bilateral venography (e.g. amputation of 1 leg, allergy to contrast media)
* Ongoing anticoagulant therapy (e.g. warfarin, heparins and Factor Xa inhibitors other than study medication) that cannot be stopped (in the opinion of the investigator/sub investigator)
* Subjects for whom epidural catheters are expected to be left in for longer than 18 hours post-operatively
* Planned intermittent pneumatic compression during treatment period.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2010-10; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
A composite endpoint of any deep vein thrombosis (proximal and/or distal), non-fatal pulmonary embolism and death from all causes | up to Day 13 (±2 days)
Treatment-emergent bleeding (major, non-major clinically relevant, other non-major) | from the first intake of study medication to no later than 2 days after the last intake of study drug

SECONDARY OUTCOMES:
deep vein thrombosis (total, proximal, distal) | up to Day 13 (±2 days)
symptomatic venous thromboembolism | up to Day 13 (±2 days)
major venous thromboembolism (proximal deep vein thromboembolism, pulmonary embolism or venous thromboembolism-related death) | up to Day 13 (±2 days)
symptomatic venous thromboembolism | within 30 days after stop of treatment with study drug

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (30):
- Japan (30):
  - Nagoya, Aichi-ken
  - Matsudo, Chiba
  - Matsuyama, Ehime
  - Fukuoka, Fukuoka
  - Kawanuma, Fukushima
  - Kōriyama, Fukushima
  - Asahikawa, Hokkaido
  - Hakodate, Hokkaido
  - Sapporo, Hokkaido
  - Kakogawa, Hyōgo
  - Kobe, Hyōgo
  - Nishinomiya, Hyōgo
  - Tsukuba, Ibaraki
  - Kyoto, Kyoto
  - Iida, Nagano
  - Sasebo, Nagasaki
  - Tomigusuku, Okinawa
  - Hirakata, Osaka
  - Izumi, Osaka
  - Izumisano, Osaka
  - Kishiwada, Osaka
  - Osaka, Osaka
  - Sakai, Osaka
  - Sayama, Osaka
  - Takatsuki, Osaka
  - Saga, Saga-ken
  - Saitama, Saitama
  - Adachi City, Tokyo
  - Nerima-ku, Tokyo
  - Toyama, Toyama